CLINICAL TRIAL: NCT00819039
Title: A Multi-center, 2-Part Study to Evaluate the Pharmacokinetics Safety and Tolerability of Aprepitant in Pediatric Patients Undergoing Surgery
Brief Title: A Study of Aprepitant (MK-0869) in Pediatric Participants Undergoing Surgery (MK-0869-148)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0869-148; 2008_569 (Other: Merck); 2008-003178-17 (EudraCT Number)
Record Dates: First submitted 2009-01-07; First posted 2009-01-08 (Estimated); Results first posted 2014-02-14 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Aprepitant; Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1: Oral Aprepitant (Experimental): In Study Part 1, participants aged 6 months to 17 years received a single oral dose of aprepitant on Day 1.
  Interventions: Drug: Aprepitant
- Part 2: Oral Aprepitant (Experimental): In Study Part 2, participants aged 6 months to 17 years received a single oral dose of aprepitant on Day 1.
  Interventions: Drug: Aprepitant
- Part 2: Intravenous Ondansetron (Active Comparator): In Study Part 2, participants aged 6 months to 17 years received a single intravenous dose of ondansetron on Day 1.
  Interventions: Drug: Ondansetron

INTERVENTIONS:
Drug: Aprepitant — Aprepitant administered orally or intraveously.
  Other Names: Emend
  Arms: Part 1: Oral Aprepitant; Part 2: Oral Aprepitant
Drug: Ondansetron — Ondansetron administered intravenously.
  Other Names: Zofran
  Arms: Part 2: Intravenous Ondansetron

SUMMARY:
This two part study will determine the appropriate dosing regimen of aprepitant for the prevention of postoperative nausea and vomiting (PONV) in pediatric participants 6 months to 17 years of age, by assessing pharmacokinetic parameters and monitoring safety and tolerability of administered doses. Part I will be an open label investigation of a single dose of aprepitant measuring pharmacokinetics at specified time points up to 48 hours after aprepitant dosing. Part II will be a double blind trial of participants randomized to receive either aprepitant or ondansetron.

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled to have surgery requiring a 48 hour (Part I) or 24 hour (Part II) hospital stay
* Participant is scheduled to receive general anesthesia
* Participant is scheduled to receive opioids (e.g. morphine or fentanyl)
* Female participants of childbearing potential must have negative pregnancy test prior to drug administration
* A female participant who is of reproductive potential must agree to remain abstinent or use a barrier form of contraception for at least 14 days prior to, throughout, and for at least one month following the last dose of study medication
* Participant weighs 6 kg or more

Exclusion Criteria:

* Participant is undergoing surgery for a life-threatening condition
* Participant is pregnant or breast feeding
* Participant has vomited within 24 hours prior to surgery
* Participant has a known history of QT prolongation or is currently taking other medicinal products that lead to QT prolongation
* Participant has an active infection (e.g., pneumonia), congestive heart failure, bradyarrythmia, any uncontrolled disease (e.g., diabetic ketoacidosis, gastrointestinal obstruction), evidence of any clinically significant respiratory, metabolic, hepatic, renal dysfunction, or a history of any illness, including morbid obesity, that might pose unwarranted risk

Ages: 6 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2009-01-26 (Actual); Primary Completion 2013-03-12 (Actual); Study Completion 2013-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC
Locations (6):
- United States (2):
  - Call for Information (Investigational Site 0003), Louisville, Kentucky
  - Call for Information (Investigational Site 0022), Nashville, Tennessee
- MSD, São Paulo, São Paulo, Brazil
- MSD, Mexico City, Mexico
- Merck Sharp and Dohme de Espana S.A., Madrid, Spain
- Merck Sharp & Dohme Ilaclari Ltd. Sti, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Chain A, Wrishko R, Vasilinin G, Mouksassi S. Modeling and Simulation Analysis of Aprepitant Pharmacokinetics in Pediatric Patients With Postoperative or Chemotherapy-Induced Nausea and Vomiting. J Pediatr Pharmacol Ther. 2020;25(6):528-539. doi: 10.5863/1551-6776-25.6.528. PMID 32839657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was conducted at 18 trial centers: 2 in Brazil, 1 in Finland, 1 in Russia, 1 in Mexico, 4 in Spain, 6 in Turkey, and 3 in the United States.
Groups:
- Part 1: Oral Aprepitant: In Study Part 1, participants aged 6 months to 17 years received a single oral dose of aprepitant for the treatment of post-operative nausea and vomiting (PONV) on Day 1.
- Part 2: Oral Aprepitant: In Study Part 2, participants aged 6 months to 17 years received a single oral dose of aprepitant for the treatment of post-operative nausea and vomiting (PONV) on Day 1.
- Part 2: Intravenous Ondansetron: In Study Part 2, particpants aged 6 months to 17 years received a single intravenous dose of ondansetron for the treatment of post-operative nausea and vomiting (PONV) on Day 1.
Period: Overall Study
Arm/Group | Part 1: Oral Aprepitant | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron
Started | 46 | 27 | 25
Completed | 44 | 27 | 24
Not Completed | 2 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Oral Aprepitant | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron | Total
Number analyzed (Participants) | 46 | 27 | 25 | 98
Age, Customized [Number; unit: Participants]
  0.5 to <2 years | 14 | 8 | 5 | 27
  2 to <6 years | 11 | 7 | 7 | 25
  6 to <12 years | 11 | 5 | 6 | 22
  12 to 17 years | 10 | 7 | 7 | 24
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 6 | 12 | 31
  Male | 33 | 21 | 13 | 67

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Curve From 0-48 (AUC0-48) of Aprepitant Following a Single Oral Dose in Study Part 1
Description: Blood samples of 0.5 mL were collected from participants for the analysis of AUC0-48 at specified time points: pre-dose, and 1, 2, 3, 4, 8, 12, 24, and 48 hours post aprepitant single dose.
Time Frame: Pre-dose, and 1, 2, 3, 4, 8, 12, 24, and 48 hours post-dose
Population: The population consisted of all participants that received at least one dose of study medication and for which AUC0-48 data were available.
Measure: Mean (Standard Deviation); unit: hr*ug/ml
Arm/Group | Part 1: Oral Aprepitant
Number analyzed (Participants) | 43
hr*ug/ml
  6 months to <2 years (n=11) | 5.97 (4.44)
  2 years to <6 years (n=11) | 4.76 (3.55)
  6 years to <12 years (n=11) | 6.16 (2.27)
  12 years to 17 years (n=10) | 6.01 (2.53)

2. Primary Outcome: Maximum Plasma Concentration (Cmax) of Aprepitant Following a Single Oral Dose in Study Part 1
Description: Blood samples were collected from participants for the analysis of Cmax up to 48 hours after dosing.
Time Frame: 48 Hours Post-Dose
Population: The population consisted of all participants that received at least one dose of study medication and for which Cmax data were available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Oral Aprepitant
Number analyzed (Participants) | 43
ng/mL
  6 months to <2 years (n=11) | 715 (445)
  2 years to <6 years (n=11) | 586 (462)
  6 years to <12 years (n=11) | 913 (294)
  12 years to 17 years (n=10) | 520 (230)

3. Primary Outcome: Time to Maximum Plasma Concentration (Tmax) of Aprepitant Following a Single Oral Dose in Study Part 1
Description: Blood samples were collected from participants for the analysis of Tmax up to 48 hours after dosing.
Time Frame: 48 Hours Post-Dose
Population: The population consisted of all participants that received at least one dose of study medication and for which Tmax data were available.
Measure: Median (Full Range); unit: Hours
Arm/Group | Part 1: Oral Aprepitant
Number analyzed (Participants) | 43
Hours
  6 months to <2 years (n=11) | 3.00 [1.00 to 8.00]
  2 years to <6 years (n=11) | 3.00 [1.03 to 12.00]
  6 years to <12 years (n=11) | 2.00 [1.00 to 8.00]
  12 years to 17 years (n=10) | 3.50 [1.00 to 11.98]

4. Primary Outcome: Plasma Concentration of Aprepitant at 24 Hours (C24 hr) Following a Single Oral Dose in Study Part 1
Description: Blood samples were collected from participants for the analysis of C24 hr at 24 hours after dosing. N/A indicates that >50% of measurements were below the lower level of quantitaion (LLOQ).
Time Frame: 24 Hours Post-Dose
Population: The population consisted of all participants that received at least one dose of study medication and for which C24 hr data were available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Oral Aprepitant
Number analyzed (Participants) | 43
ng/mL
  6 months to <2 years (n=11) | 31.0 (39.5)
  2 years to <6 years (n=11) | 58.6 (54.3)
  6 years to <12 years (n=11) | 51.1 (35.6)
  12 years to 17 years (n=10) | 81.1 (59.8)

5. Primary Outcome: Plasma Concentration of Aprepitant at 48 Hours (C48 hr) Following a Single Oral Dose in Study Part 1
Description: The mean plasma concentration of aprepitant was evaluated in participants at 48 hours following a single oral dose.
Time Frame: 48 Hours Post-Dose
Population: The population consisted of all participants that received at least one dose of study medication and for which C48 hr data were available.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Oral Aprepitant
Number analyzed (Participants) | 10
ng/mL
  6 months to <2 years (n=11) | NA (NA) — Data are not reported since >50% of the measurements were below the lower limit of quantitation (LLOQ).
  2 years to <6 years (n=11) | NA (NA) — Data are not reported since >50% of the measurements were below the lower limit of quantitation (LLOQ).
  6 years to <12 years (n=11) | NA (NA) — Data are not reported since >50% of the measurements were below the lower limit of quantitation (LLOQ).
  12 years to 17 years (n=10) | 7.25 (8.90)

6. Primary Outcome: Number of Participants Experiencing Adverse Events (AEs)
Time Frame: Up to 21 Days Post-Surgery
Population: The population consists of all participants that received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Part 1: Oral Aprepitant | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron
Number analyzed (Participants) | 46 | 27 | 25
Participants | 20 | 12 | 7

7. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to AEs
Time Frame: Day 1
Population: The population consists of all participants that received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Part 1: Oral Aprepitant | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron
Number analyzed (Participants) | 46 | 27 | 25
Participants | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With No Vomiting Up to 24 Hours Following Surgery in Study Part 2
Time Frame: Up to 24 Hours
Population: The Full Analysis Set (FAS) population was used for all efficacy evaluations and included those participants who received a full dose of active study therapy, had surgery, and had at least one post-treatment efficacy assessment.
Measure: Number; unit: Participants
Arm/Group | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron
Number analyzed (Participants) | 25 | 25
Participants | 20 | 20

9. Secondary Outcome: Number of Participants With Complete Response Up to 24 Hours Following Surgery in Study Part 2
Description: Complete response was defined as no vomiting and no use of rescue medication in 0-24 hours post-surgery.
Time Frame: Up to 24 Hours
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron
Number analyzed (Participants) | 25 | 25
Participants | 19 | 20

10. Secondary Outcome: Number of Participants With No Vomiting Up to 48 Hours Following Surgery Ini Study Part 2
Time Frame: Up to 48 Hours
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron
Number analyzed (Participants) | 25 | 25
Participants | 18 | 20

11. Secondary Outcome: Number of Participants With Complete Response Up to 48 Hours Following Surgery in Study Part 2
Description: Complete response was defined as no vomiting and no use of rescue medication in 0-48 hours post-surgery.
Time Frame: Up to 48 Hours
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron
Number analyzed (Participants) | 25 | 25
Participants | 17 | 20

12. Secondary Outcome: Number of Participants With Vomiting Frequency in Study Part 2
Time Frame: Up to 24 Hours
Population: as for outcome 8
Measure: Number; unit: Participants
Arm/Group | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron
Number analyzed (Participants) | 25 | 25
Participants
  No Vomiting | 20 | 20
  1 Vomiting Episode | 5 | 3
  2 Vomiting Episodes | 0 | 1
  3 Vomiting Episodes | 0 | 0
  >3 Vomiting Episodes | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to Day 21 post-surgery.
Description: The population consisted of all study participants that received at least one dose of study drug.
Arm/Group | Part 1: Oral Aprepitant | Part 2: Oral Aprepitant | Part 2: Intravenous Ondansetron
Serious Adverse Events (participants affected / at risk) | 3/46 | 2/27 | 0/25
Other Adverse Events (participants affected / at risk) | 14/46 | 5/27 | 4/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Oral Aprepitant (N=46) | Part 2: Oral Aprepitant (N=27) | Part 2: Intravenous Ondansetron (N=25)
Incision Site Infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anastomotic Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Oral Aprepitant (N=46) | Part 2: Oral Aprepitant (N=27) | Part 2: Intravenous Ondansetron (N=25)
Abdominal Pain (Gastrointestinal disorders) | 3 (4) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (6) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 10 (20) | 1 (5) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission.